CLINICAL TRIAL: NCT01529658
Title: A Randomized Controlled Trial of Renal Hypothermia During Partial Nephrectomy
Brief Title: Renal Hypothermia During Partial Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-767; CIHR MOP 269009
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Renal Impairment; Kidney Diseases; Urologic Diseases; Cancer; Hypothermia; Kidney Cancer
Keywords: Renal function; Renal hypothermia; Nephrology; Nephrectomy; Renal tumor; Urology; Kidney
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Urologic Diseases; Neoplasms; Hypothermia; Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Ice

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No hypothermia (No Intervention): After clamping of the renal vessels, no ice slush will be used.
- Hypothermia (Experimental): saline ice slush around kidney for 10 minutes.
  Interventions: Procedure: Renal hypothermia

INTERVENTIONS:
Procedure: Renal hypothermia — Within 10 seconds of clamping the renal vessels, the kidney will be encased with saline ice slush for a period of 10 minutes. The slush will be created from sterile saline using an operating room slush machine. The slush is applied by the surgeon and lightly packed around the kidney to ensure complete coverage with at least a 2 cm layer. Slush removal is performed by the surgeon beginning at the 10 minute mark. Enough slush is removed to uncover the tumour area. Surgical incision of the kidney begins as soon as the tumour area is uncovered.
  When reconstruction of the kidney is complete, the slush is completely removed from the surgical field and the clamps are removed from the renal vein and artery.
  Other Names: Ice
  Arms: Hypothermia

SUMMARY:
The Objective is to determine if renal hypothermia during open partial nephrectomy results in improved post-operative renal function compared to warm ischemia.

Primary Aim is to determine the effect of hypothermia on preservation of overall renal function compared to no hypothermia in patients who require hilar vessel clamping during open partial nephrectomy for a renal tumor.

Hypothesis: Hypothermia will result in improved post-operative preservation of overall renal function.

Secondary Aim is to determine the effect of hypothermia on preservation of affected renal function (kidney with the tumor) compared to no hypothermia in patients who require hilar vessel clamping during open partial nephrectomy for a renal tumor.

Hypothesis: Hypothermia will result in improved post-operative preservation of affected renal function.

DETAILED DESCRIPTION:
The incidence of renal cell carcinoma is increasing and in 2008 it is estimated that over 51,000 new renal cancers will be diagnosed in the United States. To preserve renal function, urologists commonly remove the diseased segment of the kidney (partial nephrectomy) instead of removing the entire kidney (radical nephrectomy). While the benefit of preserving function in patients with renal cell carcinoma has become clear, optimal preservation techniques are yet to be determined. Specifically, the role of hypothermia during partial nephrectomy has been inadequately studied despite theoretical benefit. The investigators objective is to assess the effectiveness of renal hypothermia during partial nephrectomy. The investigators hypothesis is that renal hypothermia during partial nephrectomy results in improved post-operative renal function compared to warm ischemia.

Methods: To test the investigators hypothesis, 180 partial nephrectomy patients will be randomized to cold or warm ischemia. Global and side-specific renal function will be assessed pre-operatively and 12 months post-operatively using radionucleotide clearance and renal scintigraphy.

Significance: To the investigators knowledge, this study will be the first prospective trial to evaluate the clinical impact of renal hypothermia during partial nephrectomy. Since renal function preservation is the primary purpose of partial nephrectomy, these findings will have an important impact on surgical technique and patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with a renal mass deemed amenable to an open partial nephrectomy regardless of stage, histology, presence of solitary kidney, multiple tumors or renal function. Participating surgeons will identify patients they consider to be appropriate candidates for partial nephrectomy with or without renal hypothermia.
* Willing to consent to randomization
* Willing to comply with study protocol

Exclusion Criteria:

* Bilateral renal tumours with planned surgery either partial or radical nephrectomy on the contralateral kidney within the 12 months of the study.
* Life expectancy < 3 months as deemed by treating physician
* Age less than 18 years old
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2012-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Renal function | 12 months
  Glomerular filtration rate will be measured using the plasma clearance of 99mTc-DTPA.

SECONDARY OUTCOMES:
Difference in affected renal function | 12 months
  Side-specific renal function will be calculated by the product of overall glomerular filtration (determined from 99mTc-DTPA plasma clearance) and relative renal contribution (determined from 99mTc-DTPA renal scintigraphy).

CONTACTS AND LOCATIONS:
Overall Officials: Ilias Cagiannos, MD, Principal Investigator — The Ottawa Hospital, Ottawa Hospital Research Institute
Locations (6):
- Canada (6):
  - Capital Disctrict Health Authority, Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - London Health Science Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Centre hospitalier universitaire de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breau RH, Cagiannos I, Knoll G, Morash C, Cnossen S, Lavallee LT, Mallick R, Finelli A, Jewett M, Leibovich BC, Cook J, LeBel L, Kapoor A, Pouliot F, Izawa J, Rendon R, Fergusson DA. Renal hypothermia during partial nephrectomy for patients with renal tumours: a randomised controlled clinical trial protocol. BMJ Open. 2019 Jan 3;9(1):e025662. doi: 10.1136/bmjopen-2018-025662. PMID 30610026